CLINICAL TRIAL: NCT05088655
Title: Bioequivalence Study of Different Formulations of Hetrombopag Olamine Tablets in Healthy Subjects
Brief Title: A Bioequivalence Study of Hetrombopag in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR8735-114
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Sever Aplastic Anaemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: T - R- R (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet
- Treatment group B: R -T - R (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet
- Treatment group C: R- R-T (Experimental)
  Interventions: Drug: Hetrombopag Olamine Tablet

INTERVENTIONS:
Drug: Hetrombopag Olamine Tablet — Hetrombopag Olamine Tablet (T: test formulation) Hetrombopag Olamine Tablet (R: reference formulation)

SUMMARY:
This study consists of two parts. Part 1 is a pilot BE study, and Part 2 is a pivotal study to demonstrate the bioequivalence of test and reference formulation, both of which adopt a single-center, randomized, open-label, three-period crossover design.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);

Exclusion Criteria:

1. Allergic constitution;
2. History of drug use, or drug abuse screening positive;
3. Alcoholic or often drinkers;
4. History of deep vein thrombosis, or any other thromboembolic event;
5. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 0-120 hours post dose
Area Under the plasma concentration vs time curve (AUC0-120) | 0-120 hours post dose
area under the plasma concentration vs time curve (AUC0-inf) | 0-infinity

SECONDARY OUTCOMES:
Time to Reach Maximum Drug Concentration in Plasma After Single Dose (Tmax) | 0-120 hours post dose
Half-life Associated With the Terminal Slope (t½) | 0-120 hours post dose
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 26

CONTACTS AND LOCATIONS:
Locations (1):
- The People's Hospital Of Liaoning Province, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided